CLINICAL TRIAL: NCT02199717
Title: An Institutional Pilot Study to Investigate Physical Activity Patterns in Boys With Hemophilia
Acronym: HEPS
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Hemophilia Society (Other)
Responsible Party: Principal Investigator, Vanessa Bouskill, Nurse Practitioner, The Hospital for Sick Children
Other Study IDs: 1000039947
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Hemophilia A; Hemophilia B; Factor VIII Deficiency; Factor IX Deficiency
Keywords: Physical Activity; Accelerometer; Exercise; Obesity; BMI
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Motor Activity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Boys with Hemophilia: Accelerometer use for 1 week.
  Interventions: Device: Accelerometer

INTERVENTIONS:
Device: Accelerometer
  Other Names: ActiLife; Kinesoft

SUMMARY:
This pilot project was developed to investigate subjective and objective data related to the patterns of physical activity participation among hemophilia patients (FVIII or FIX) between the ages of 5 and 18 years. Physical activity participation among different levels of disease severity will be compared using accelerometers to calculate the amount of time spent in moderate to vigorous physical activity (MVPA) and the number of bouts of MVPA; additionally, data will be collected from two validated questionnaires (PedHAL and 3 day physical activity recall). Current literature that relates level of physical activity to disease severity in the pediatric hemophilia population is limited. The information gained about the type and quantity of physical activity participation in children with varying levels of hemophilia will assist in the development of education and interventions to promote good physical activity and potentially examine the role of tailored prophylaxis.

DETAILED DESCRIPTION:
Objectives:

1. To determine if the amount of time spent performing moderate to vigorous physical activity (MVPA) and the number of bouts of MVPA engaged in on a weekly basis differs by the level of disease severity in the pediatric hemophilia population.
2. To determine if recorded physical activities and intensity of activities from self-report questionnaires (PedHAL and 3 day physical activity recall - 3DPAR) differ according to the severity of hemophilia.
3. To determine if, among patients with hemophilia, there is a relationship between physical activity level and patient age, weight, and body mass index (BMI).

Specific Aims:

•Aim # 1: The primary aim of the study is to determine if there are differences in the amount of time spent in MVPA by level of disease severity of children with hemophilia.

Secondary Aims:

* Aim # 2: To determine if there are meaningful differences in the accumulation of MVPA (bouts of exercise) by disease severity of children with hemophilia.
* Aim # 3: The compare the findings from Aim #1 and #2 to the NHANES (National Health and Nutrition Examination Survey) data, recognizing that this survey provides a comparative healthy normal cohort.
* Aim # 4: To investigate MVPA with these data collected from the PedHAL (11) and the 3DPAR (12) by disease severity of children with hemophilia.
* Aim # 5: The review and determine the relationship between physical activity participation and timing of prophylaxis factor replacement and whether participation is limited to days of factor infusion.
* Aim #6: To investigate the amount of physical activity and how it relates to age, weight, and patient body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* 5-17 years of age, has a diagnosis of Hemophilia A or B.

Exclusion Criteria:

* Muscle or joint bleed within 4 weeks of study.
* Pre-existing co-morbidities that would affect physical activity participation.
* Unable to cooperate with study protocol.
* Unable to speak, read, or understand English.

Ages: 5 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be 5 to 18 years of age with a diagnosis of hemophilia with no history of inhibitors or pre-existing co-morbidity (e.g. cerebral palsy, chronic respiratory conditions, congenital heart defects) that can affect activity participation.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Bouskill, NP, MN, Principal Investigator — The Hospital for Sick Children
Locations (1):
- SickKids, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Boys With Hemophilia: Use of accelerometer for 1 week
Period: Overall Study
Arm/Group | Boys With Hemophilia
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 42 boys with severe hemophilia 24 boys with moderate/mild hemophilia
Arm/Group | Boys With Hemophilia
Number analyzed (Participants) | 66
Age, Customized [Number; unit: participants]
  <=18 years | 66
  Between 18 and 65 years | 0
  >=65 years | 0
Sex/Gender, Customized [Number; unit: Participants] — All male
  Participants
    Female | 0
    Male | 66
Region of Enrollment [Number; unit: participants] — SickKids catchment area
  participants
    Canada | 66
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: BMI was grouped by hemophilia severity.
  kg/m2
    Severe Hemophilia: number analyzed (Participants) | 42
    Severe Hemophilia | 20.05 (5.82)
    Mild/Moderate Hemophilia: number analyzed (Participants) | 24
    Mild/Moderate Hemophilia | 21.93 (5.34)
On demand or Prophylaxis Regimen [Count of Participants; unit: Participants] — On demand (only treated for bleeds) Prophylaxis (treated to prevent bleeds from occuring) Population: Grouped by hemophilia severity.
  Participants
    Severe Hemophilia: number analyzed (Participants) | 42
    Severe Hemophilia: On prophylaxis | 42
    Severe Hemophilia: On demand | 0
    Mild/Moderate Hemophilia: number analyzed (Participants) | 24
    Mild/Moderate Hemophilia: On prophylaxis | 5
    Mild/Moderate Hemophilia: On demand | 19
Severity of Hemophilia [Count of Participants; unit: Participants] — Severe <1% FVIII (Factor 8 Deficiency/Hemophilia A) or FIX (Factor 9 Deficiency/Hemophilia B) Moderate/Mild >1% FVIII or FIX
  Participants
    Severe | 42
    Mild/Moderate | 24

OUTCOME MEASURES:

1. Primary Outcome: MVPA
Description: To determine if the amount of time spent performing moderate to vigorous physical activity (MVPA) engaged in on a weekly basis differs by the level of disease severity in the pediatric hemophilia population.
Time Frame: 7 days
Population: All statistical analyses were completed using SAS 9.4 (SAS Institute Inc., Cary, NC, USA). Descriptive statistics such as mean (± SD) and range were calculated and provided for demographic variables, accelerometry variables and questionnaire outcomes. Differences between the two groups were examined in exploratory analyses.
Measure: Mean (Standard Deviation); unit: minutes per day
Groups:
- Severe Hemophilia: Severe Hemophilia
- Mild/Moderate Hemophilia: Mild/Moderate Hemophilia
Arm/Group | Severe Hemophilia | Mild/Moderate Hemophilia
Number analyzed (Participants) | 42 | 24
minutes per day | 48 (20) | 55 (18)
Statistical Analysis 1: Comparison: Severe Hemophilia; All statistical analyses were completed using SAS 9.4 (SAS Institute Inc., Cary, NC, USA). Descriptive statistics such as mean (± SD) and range were calculated and provided for demographic variables, accelerometry variables and questionnaire outcomes. Differences between the two groups (mild/moderate versus severe haemophilia) were examined in exploratory analyses; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Sedentary Time
Description: To determine if the amount of time spent in sedentary time on a weekly basis differs by the level of disease severity in the pediatric hemophilia population.
Time Frame: 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Severe Hemophilia | Mild/Moderate Hemophilia
Number analyzed (Participants) | 42 | 24
minutes per day | 633.4 (121.3) | 327 (78.73)
Statistical Analysis 1: Comparison: Severe Hemophilia vs Mild/Moderate Hemophilia; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 306.4, 95% CI 2-sided [254.8 to 358]

ADVERSE EVENTS:
Time Frame: Adverse events were documented for the duration of study for each participant (duration being 1 week).
Arm/Group | Severe Hemophilia
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No